CLINICAL TRIAL: NCT04024761
Title: A Phase 1 Trial of CIML NK Cell Infusion for Myeloid Disease Relapse After Hematopoietic Cell Transplantation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Principal Investigator, Roman Shapiro, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-265
Record Dates: First submitted 2019-07-17; First posted 2019-07-18 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-02

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes; Myeloproliferative Neoplasm; Juvenile Myelomonocytic Leukemia
Keywords: Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Myeloproliferative Disorders; Leukemia, Myelomonocytic, Juvenile; Leukemia | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CIML NK (Experimental): * CIML NK cells will be administered intravenously on day 0.
  * Fludarabine will be administered as IV infusion once daily for 3 doses beginning on day -5.
  * Cyclophosphamide will be administered as IV infusion on days -5 and -4.
  Interventions: Biological: CIML NK; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: CIML NK — CIML NK cells have enhanced ability to recognize and kill leukemia targets
Drug: Fludarabine — Fludarabine is a chemotherapy agent
Drug: Cyclophosphamide — Cyclophosphamide (CP), also known as cytophosphane among other names, is a chemotherapy agent

SUMMARY:
This research study is studying cytokine induced memory-like natural killer (CIML NK) cells combined with IL-2 in adult patients (18 years of age or older) with Acute Myeloid Leukemia (AML), Myelodysplastic Syndrome (MDS) and Myeloproliferative Neoplasms (MPN) who relapse after haploidentical hematopoietic cell transplantation (haplo-HCT) or HLA matched stem cells. This study will also study CIML NK cell infusion combined with IL-2 in pediatric patients (12 years of age or older) with AML, MDS, JMML who relapse after stem cell transplantation using HLA-matched related donor or related donor haploidentical stem cells.

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies. "Investigational" means that the intervention is being studied.

The U.S. Food and Drug Administration (FDA) has not approved CIML NK Cell Infusion as a treatment for relapsed disease.

ELIGIBILITY:
1. Inclusion Criteria:

   1.1 Relapse or post-transplant persistence of AML, MDS (including JMML) or MPN (CMML, myelofibrosis or MDS/MPN). Disease relapse or persistence will be defined as any measurable disease by morphology, flow-cytometry, validated tests for minimal residual disease or disease-defining mutations in the bone marrow, or non-immune privileged extramedullary sites.

   1.2 Persistence of disease within 4 weeks before planned NK cell infusion and at least 2 weeks after completion of immune suppression taper as long as it is > 2 months after stem cell transplantation for both adult and pediatric patients. If 2 weeks after completion of the immune suppression taper is still within 2 months of the most recent stem cell transplant, then chemotherapy with Fludarabine/Cyclophosphamide would need to start no earlier than at least 2 months after the transplant. For adults, disease persistence after a second transplant is allowed as long as the most recent transplant was a haploidentical or HLA matched stem cell transplant. In the pediatric cohort, disease persistence or recurrence after a second transplant is allowed as long as the most recent transplant was a haploidentical or matched related donor SCT.

   1.3 Available original donor (same donor as used for the most recent haploidentical or HLA matched stem cell transplant for adults, or for the most recent matched related donor or related haploidentical donor for pediatrics) that is willing and eligible for non-mobilized collection.

   1.4 Age ≥12 years.

   1.5 ECOG performance status ≤2. For For patients in the pediatric cohort, this corresponds to a Lansky (patients <16 years) or Karnofsky (≥16years) performance status of ≥50.

   1.6 T cell chimerism ≥20% donor-derived within the 4 weeks prior to cell infusion.

   1.7 Patient with ≤80% bone marrow involvement within 4 weeks prior to cell infusion. Medications like hydroxyurea, decitabine or cytarabine are allowed to control rising blasts between study enrollment and cell infusion.

   1.8 No systemic corticosteroid therapy for GVHD (≤ 5mg of prednisone or equivalent dose of systemic steroids for non-GVHD, non-autoimmune indications are allowed) for at least 4 weeks prior to cell infusion. Patients on systemic GVHD prophylaxis medications such as tacrolimus or sirolimus need to be off these medications for at least 4 weeks prior to cell infusion.

   1.9 No other systemic medications/treatments (e.g. ECP) for GVHD for at least 4 weeks prior to cell infusion.

   1.10 Ability of the patient or legal guardian to understand and the willingness to sign a written informed consent document.

   1.11 Adequate organ function within 2 weeks of NK cell infusion as defined below:
   * Total bilirubin: ≤1.5 x institutional upper limit of normal (ULN) (except Gilbert's or disease-related hemolysis, then <3 x ULN)
   * AST(SGOT)/ALT(SGPT): ≤3 x institutional ULN
   * Serum creatinine ≤2.0mg/dL
   * O2 saturation: ≥90% on room air
   * LVEF >40%. If there is no clinical evidence of a change in cardiovascular function from the time of pre-transplantation ECHO, then there is no need to repeat it. Otherwise, an ECHO will need to be repeated within 2 weeks of NK cell infusion.

   1.12 Negative pregnancy test for women of childbearing potential only.

   1.13 The effects of CIML NK cells and IL-2 on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after the last IL-2 dose administration.
2. Exclusion Criteria:

2.1 Extramedullary relapse involving immuno-privileged sites (e.g. CNS, testes, eyes). Other sites of extramedullary relapse (e.g. leukemia cutis, granulocytic sarcoma) are acceptable.

2.2 Participants who have had investigational agents within 4 weeks prior to cell infusion (6 weeks for nitrosoureas or mitomycin C), or immunotherapy within 8 weeks prior, or those who have not recovered from adverse events due to agents administered more than 4 weeks prior or standard chemotherapy administered more than 14 days ago. Use of hydroxyurea, hypomethylating agents, low-dose cytarabine or venetoclax to control counts within 4 weeks prior to cell infusion is permitted with study PI approval but would need to be stopped 1 day prior to administration of Fludarabine and Cyclophosphamide preceding the NK cell infusion (provided that there are no ongoing AEs attributed to these agents that would preclude start of lymphodepletion in the view of the investigator). Patients on standard of care FLT-3, IDH1, and IDH2 inhibitors can stay on this treatment. Therapy with BCR-ABL inhibitors or bcl-2 inhibitors must be stopped 2 weeks before NK cell infusion and may be resumed after the end of the DLT period.

2.3 Prior history of Donor Lymphocyte Infusion (DLI) within 8 weeks of CIML NK infusion. DLI that was given before this time period and that did not result in any GVHD requiring systemic treatment is not an exclusion criterion.

2.4 Prior history of severe (grade 3 or 4) acute GVHD, or ongoing active GVHD requiring systemic treatment.

2.5 Solid organ transplant recipient. Prior allogeneic HLA matched or mismatched stem cell transplant is allowed in the pediatric cohort. Prior HLA matched related donor or HLA matched unrelated donor stem cell transplant is allowed in the adult cohort.

2.6 History of allergic reactions attributed to compounds of similar chemical or biologic composition to IL-2 or other agents used in study.

2.7 Autoimmune disease: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]) and motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome and Myasthenia Gravis). Patients with Hashimoto's thyroiditis are eligible to go on study.

2.8 Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

2.9 Patients who develop a critical illness prior to NK cell infusion that would contraindicate the administration of Fludarabine and Cyclophosphamide conditioning. Patients who recover from such illness may still be eligible, but this must be reviewed with the study PI. A repeat bone marrow examination may be required depending on the timing of recovery. Patients who become critically ill on the planned day of NK cell infusion are excluded if the NK cell infusion cannot be given within 48 hours of the planned day 0.

2.10 Pregnant women are excluded from this study because of the unknown teratogenic risk of CIML NK cells and IL-2 and with the potential for teratogenic or abortifacient effects by Flu/Cy chemotherapy regimen. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with CIML NK cells and IL-2, breastfeeding should be discontinued if the mother is treated on this study.

2.11 HIV-positive participants are ineligible because of the potential for pharmacokinetic interactions with anti-retroviral agents used in this study. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy.

2.12 Individuals with active uncontrolled hepatitis B or C, HIV, or HTLV-1 are ineligible as they are at high risk of lethal treatment-related hepatotoxicity after HSCT.

2.13 Individuals with a history of a different malignancy are ineligible except for the following circumstances: 1. History of other malignancy and have had complete remission of disease for at least 2 years; 2. Diagnosed and treated within the past 2 years for: nonmetastatic melanoma, surgically resected (not needing systemic chemotherapy) squamous cell carcinoma of skin and nonmetastatic prostate cancer not needing systemic chemotherapy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-08-31 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety | 6 Weeks
  To determine the maximum tolerated dose (MTD) of CIML NK cell infusion followed by low-dose IL-2

SECONDARY OUTCOMES:
ORR (Objective Response Rate) | 28 days
  To determine complete remission (CR/CRi) rate after CIML NK cell infusion plus IL-2
LFS and OS | 100 Days, 1 Year
  To determine the rate of leukemia-free survival (LFS) and overall survival (OS) at day 100 and at 1 year post cell CIML NK cell infusion plus IL-2
Acute GVHD (Incidence, Severity) | 100 Days, 6 Months
  To determine the incidence and severity of acute GVHD rates after CIML NK cell infusion plus IL-2
Chronic GVHD (Incidence, Severity) | 1 Year
  To determine the incidence and severity of chronic GVHD rates after CIML NK cell infusion plus IL-2

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Baumeister, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Shapiro RM, Birch GC, Hu G, Vergara Cadavid J, Nikiforow S, Baginska J, Ali AK, Tarannum M, Sheffer M, Abdulhamid YZ, Rambaldi B, Arihara Y, Reynolds C, Halpern MS, Rodig SJ, Cullen N, Wolff JO, Pfaff KL, Lane AA, Lindsley RC, Cutler CS, Antin JH, Ho VT, Koreth J, Gooptu M, Kim HT, Malmberg KJ, Wu CJ, Chen J, Soiffer RJ, Ritz J, Romee R. Expansion, persistence, and efficacy of donor memory-like NK cells infused for posttransplant relapse. J Clin Invest. 2022 Jun 1;132(11):e154334. doi: 10.1172/JCI154334. PMID 35349491